CLINICAL TRIAL: NCT05496218
Title: Metabolomic Profile in Women With and Without Endometriosis: a Case-control Study
Brief Title: Metabolomic Profile in Women With and Without Endometriosis
Acronym: METABOLENDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0009220 U
Record Dates: First submitted 2022-03-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis; Endometriosis-related Pain; Infertility
Keywords: Metabolomics; Personalized medicine; Diagnosis
MeSH Terms: conditions — Endometriosis; Infertility; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Single-center case-control study.
Masking Description: Study participants will be subjected to blood sampling that is not part of the routine clinical practice, so it's an interventional study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis group (Experimental): Endometriosis group are women aged 18-45 with a histologically confirmed diagnosis of endometriosis. At study entry, we will collect morning blood samples.
  Interventions: Diagnostic Test: Blood samples
- Control Group (Experimental): Control group are women aged 18-45 surgically verified not to have endometriosis. At study entry, we will collect morning blood samples.
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — At study entry, we will collect morning blood samples from fasting women. participants will be asked with an interview on demographic and lifestyle characteristics, health-related behaviours, the existence and duration of infertility, medical history, and history of hormonal or surgical treatments for endometriosis. Pain symptoms before surgery will be evaluated through a 10 cm long one-dimensional visual-analogue scale (VAS). In addition, women will be asked to report about their usual weekly food consumption in the previous year. Information on the diet will be based on a reproducible and valid food frequency questionnaire. Energy and mineral and macro-and micronutrient intakes will be estimated using the most recent update of an Italian Food Consumption Database.

SUMMARY:
The pathogenesis of endometriosis is very complex as several factors, including genetic, environmental and lifestyle-related factors, are involved in the development, progression and maintenance of the disease. In particular, there are emerging evidences that prostaglandin metabolism, chronic inflammatory processes and circulating estrogen levels are involved in the pathogenesis of endometriosis. Pelvic pain, in particular dysmenorrhea, is the most typical symptom caused by the production of prostaglandins and pain mediators associated with the peritoneal inflammatory state.

Metabolomics strives to measure all metabolites, such as sugars, amino acids, acylcarnitines, organic acids, and lipids, present in a given biological sample. Thus, metabolomics represents a reflection of phenotypic changes in an organism in response to the presence of a certain disease, genetic changes, and nutritional, toxicological, environmental, and pharmacological influences, providing a means to more accurately capture exogenous exposures and evaluate endogenous biomarkers.

Regarding endometriosis, the targeted metabolomics studies focused mainly on lipids, and the non-targeted studies also identified mainly lipids, amino acids, and intermediary metabolites as the most important variables.

The combinations of metabolomics data together with clinical ones are of utmost importance in endometriosis research. This approach might lead to the construction of models/algorithms useful to better define diagnostic/prognostic characteristics of women who have endometriosis, identify environmental and modifiable risk factors, elucidate pathogenetic mechanisms, and contribute to better tailor medical treatments.

In particular, metabolomics may provide a means to capture exogenous exposures and evaluate endogenous biomarkers more accurately.

The main objective of the present research project is to evaluate potential variations in the plasma metabolomic profile of women affected by endometriosis (as compared with a control group) as a consequence of pathophysiologic alterations associated with this disorder.

Secondary objectives are:

1. to evaluate potential variations in the plasma metabolomic profile of endometriosis patients with different phenotypes of the disease: peritoneal endometriosis, ovarian endometriosis, deep infiltrating endometriosis;
2. to evaluate potential variations in the plasma metabolomic profile of endometriosis patients in relation to the presence of endometriosis-related painful symptoms and/or infertility.

There is strong evidence that endometriosis has a negative impact on women's quality of life, with severe long-term consequences and substantial social costs. Our findings might lead to the construction of models/algorithms useful to better define diagnostic/prognostic characteristics of women who have endometriosis, identify environmental and modifiable risk factors, elucidate pathogenetic mechanisms, and contribute to better tailoring medical treatments.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial glands and stroma outside the uterine cavity. It is an estrogen-dependent chronic inflammatory disease, in which the ectopic endometrium grows and proliferate under the action of estradiol, which plays a pro-inflammatory and anti-apoptotic role. Ectopic endometrium can be found on the ovaries in the pelvic peritoneum, rectovaginal septum, and other pelvic sites; this thus defines at least three different entities: peritoneal, ovarian, and deep infiltrating endometriosis. Estimates show that up to 10% of premenopausal women and 35% to 50% of women with infertility, pelvic pain or both have endometriosis. Pelvic pain, in particular dysmenorrhea, is the most typical symptom of endometriosis, caused by the production of prostaglandins and pain mediators associated with the peritoneal inflammatory state. Thus, endometriosis significantly impairs the quality of life of women, with substantial social costs. The pathogenesis of endometriosis is very complex as several factors, including genetic, environmental and lifestyle-related factors, are involved in the development, progression and maintenance of the disease. In particular, there are emerging evidences that prostaglandin metabolism, chronic inflammatory processes and circulating estrogen levels are involved in the pathogenesis of endometriosis.

Metabolomics strives to measure all metabolites, such as sugars, amino acids, acylcarnitines, organic acids, and lipids, present in a given biological sample. Metabolomics represents a reflection of phenotypic changes in an organism in response to the presence of a certain disease, genetic changes, and nutritional, toxicological, environmental, and pharmacological influences.

In particular, metabolomics may provide a means to capture exogenous exposures and evaluate endogenous biomarkers more accurately. For example, a study on nutritional metabolomics and breast cancer risk- an estrogen-dependent disease as endometriosis and that shares similar diet-related risk factors such as high intake of alcohol, red meat and low intake of fruits and vegetables - found that pre-diagnostic serum concentrations of metabolites related to alcohol, vitamin E, and animal fats were associated with estrogen receptor positive (ER+) breast cancer risk.

Regarding endometriosis, the targeted metabolomics studies focused mainly on lipids, and the non-targeted studies also identified mainly lipids, amino acids, and intermediary metabolites as the most important variables.

The combinations of metabolomics data together with clinical ones are of utmost importance in endometriosis research.

This approach might lead to the construction of models/algorithms useful to better define diagnostic/prognostic characteristics of women who have endometriosis, identify environmental and modifiable risk factors, elucidate pathogenetic mechanisms, and contribute to better tailoring medical treatments.

As preliminary evidence suggests that endometriosis causes metabolic dysregulation, the investigators hypothesize that metabolomics could represent a promising method to diagnose women with endometriosis and women without endometriosis early.

Moreover, the investigators hypothesized that the metabolic approach could represent a possible diagnostic tool that allows a better description of the disease phenotype (peritoneal, ovarian or deep infiltrating endometriosis), identifying new biomarkers and clarifying the metabolic pathways involved in the disease. In addition, this approach could represent a valuable tool to early identify women with endometriosis at risk to develop painful symptoms and/or infertility.

There is strong evidence that endometriosis has a negative impact on women's quality of life, with severe long-term consequences that should be carefully addressed in developing national healthcare programs. Our findings may lead to the implementation of more effective instruments for early diagnosis and tools for identifying environmental and modifiable risk factors, particularly in relation to nutrition, elucidating the underlying pathogenetic mechanisms.

Preliminary data:

The first metabolomics study to identify novel biomarkers of endometriosis was published in 2012. In addition, a systematic review was recently published about the contribution of metabolomics to the identification of diagnostic and prognostic biomarkers for uterine diseases, including 17 studies on endometriosis. The targeted metabolomics studies focused mainly on lipids, and the non-targeted studies also identified mainly lipids, amino acids, and intermediary metabolites as the most important variables. The highest diagnostic accuracies were reported for the plasma/serum metabolic signatures that separated healthy women from endometriosis patients. For stratification between infertile women and endometriosis patients, a panel of serum metabolites was identified in a small case/control discovery study, with a high AUC of 0.99: lactate, 2-hydroxybutyrate, succinate, and lysine, the data on this issue are however very limited.

ELIGIBILITY:
Inclusion Criteria:

1. Endometriosis group.

   * are women aged 18-45
   * histologically confirmed diagnosis of endometriosis consecutively observed at the "Endometriosis center" Fondazione IRCCS Ospedale Maggiore Policlinico, Milan.
   * Only incident cases (i.e. diagnosis within three months before study entry) will be eligible.
2. Control group are women aged 18-45 surgically verified not to have endometriosis. In this group, the indications for surgery will be abdominal surgical emergencies, tubal infertility, non-endometriotic ovarian cysts, or uterine fibroids. Controls will be identified consecutively at the same institution where cases have been identified.

Exclusion Criteria:

1. Endometriosis group:

   * the presence of diseases causing pelvic pain other than endometriosis,
   * hormonal treatment in the past two months before surgery,
   * menopausal state
   * pregnancy
   * gynecological cancers
   * pelvic inflammatory disease
2. Control group:

   * hormonal treatment in the past two months before surgery
   * menopausal state
   * pregnancy
   * gynecological cancers.
   * pelvic inflammatory disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-09 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Determination of plasma metabolomic profile using an LC-MS/MS targeted metabolomic method | 24 months
  Potential variations in the plasma metabolomic profile of endometriosis patients as a consequence of pathophysiologic alterations associated with this disorder. Metabolomic set-up will be evaluated with a targeted approach and instrumentation based on the triple quadrupole mass Spectrometry interfaced with liquid chromatography at very high pressure. Metabolomic profile analysis of subjects will be conducted using a targeted LC-MS/MS metabolomic method through the AbsoluteIDQ kit¹ p180. A good inter-laboratory reproducibility of this test was reported for measurements of the above metabolites in human plasma. The instrumentation will consist of a high pressure liquid chromatograph Agilent coupled with hybrid triple quadrupole/linear ion trap mass spectrometer with an electrospray ionization source. The test shall be conducted according to the manufacturer's instructions.

SECONDARY OUTCOMES:
Relation between Plasma metabolomic profile and endometriosis phenotypes through a questionnaire | 24 months
  We expect that women in the endometriosis group will differ with regard to metabolomic profile with respect to the disease phenotype different phenotypes of the disease: peritoneal endometriosis, ovarian endometriosis, deep infiltrating endometriosis. We will not use for this outcome no scale.
Plasma metabolomic profile and fertility in terms of pregnancy rate | 24 months
  we expect that women in the endometriosis group will differ with regard to metabolomic profile with respect the presence infertility
Relation between Plasma metabolomic profile and pelvic pain evaluated through visual-analogue scale (VAS) | 24 months
  we expect that women in the endometriosis group will differ with regard to metabolomic profile with respect the presence of endometriosis-related painful symptoms. VAS scale, from 1 meaning better outcome to 10 meaning worse outcome.
Plasma metabolomic profile and dietary exposure through food frequency questionnaire (FFQ) | 24 months
  we expect that women in the endometriosis group will differ with regard to metabolomic profile with respect the dietary exposure. to report about their usual weekly food consumption in the previous year. Information on the diet will be based on a reproducible and valid food frequency questionnaire (doi: 10.1016/j.rbmo.2020.07.011. )

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Vercellini, Prof., Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No